CLINICAL TRIAL: NCT05868876
Title: A Phase Ia/Ib Open Label，Clinical Study Evaluating the Safety, Tolerability and Preliminary Efficacy of AK127 in Combination With AK104 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK127-103
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The dose escalation stage, dose expansion stage of AK127 combination with AK104 (Experimental): The dose escalation stage： 5 dose groups were set up, which were 0.3mg/kg、1 mg/kg, 3 mg/kg, 7.5 mg/kg, 15 mg/kg Q3W in dose escalation stage; The dose expansion stage： 8 cohorts with different indications were included in each group with 10-20 subjects in dose expansion stage.
  Interventions: Drug: AK127 Q3W IV infusion ,AK104 10mg/kg Q3W IV infusion

INTERVENTIONS:
Drug: AK127 Q3W IV infusion ,AK104 10mg/kg Q3W IV infusion — AK127 is administered intravenously according to the frequency Q3W and different dosage of administration at different stages.AK104 is administered intravenously according to the frequency and dosage 10mg/kg Q3W.

SUMMARY:
A Phase Ia/Ib open label，clinical study evaluating the safety, tolerability and preliminary efficacy of AK127 in combination with AK104 in patients with advanced malignant tumors

DETAILED DESCRIPTION:
Immunocheckpoint inhibitors has greatly improved the efficacy of cancer treatment,such as in non-small cell lung cancer, melanoma, urothelial carcinoma and other tumor species, greatly improving patient survival. However, some patients still do not benefit from current immunotherapy (PD- (L) 1, or CTLA-4), suggesting that there are other mechanisms that limit the immune response within the tumor.As a result, the current immune checkpoint inhibitors (PD- (L) 1, CTLA-4) are not effective or even ineffective in some patients.

AK104 is a humanized immunoglobulin G1 (IgG1) bispecific antibody (BsAb),AK104 binds both programmed cell death 1 (PD-1) and cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) and blocks the interaction of PD-1/ programmed cell death ligand 1 (PD-L1), PD-1/PD-L2, CTLA-4/B7.1 and CTLA-4/B7.2.In June 2022, Akeso bis-specific antibody Cardonilimab (AK104) was approved by the CDE for marketing in the treatment of patients with recurrent or metastatic cervical cancer who have failed previous platinum-containing chemotherapy.

AK127 is a TIGIt-targeting IgG1 monoclonal antibody with complete Fc function. It can bind to human immune cells TIGIT with high affinity and competitively block the binding of TIGIT to its ligands CD155 and CD112.Elimination of Treg in tumor by NK cells and enhancement of anti-tumor activity of CD8+T cell , without causing regulatory T cell depletion, thus promoting anti-tumor immune response.AK127 is expected to be a more effective immune checkpoint inhibitor.

The simultaneous blocking of PD1/PDL1, CTLA4 and TIGIT is expected to simultaneously relieve tumor immunosuppression at multiple immune checkpoints, enhance anti-tumor immune response, and provide more clinical solutions. AK104 is PD1 and CTLA4 bispecific antibody, and AK127 is TIGIT monoclonal antibody.Combined application may further enhance the antitumor effect.The objective of this study was to explore the safety, tolerability, pharmacokinetics, pharmacodynamics, and initial antitumor activity of AK104 combined with AK127 in advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1.The subject must sign the written informed consent form(ICF) voluntarily. 2.Aged ≥ 18 to ≤ 75 years,male and female at the time of enrollment. 3.Eastern Cooperative Oncology Group(ECOG) performance status score of 0 or 1. 4.Life expectancy≥ 3 months. 5.Patients with histologically or cytologically confirmed advanced, recurrent, or metastatic malignancies were enrolled in the phase Ia dose escalation phase;Selected tumor species were enrolled in phase Ib dose extension.Patients with advanced metastatic malignancies who have failed first-line, or second-line, or third-line, or fourth-line standard therapies, or who not appropriate for standard treatment, cannot tolerate chemotherapy, or do not have effective standard therapies.

  6. According to RECIST v1.1, there is at least one measurable lesion, and the lesion is suitable for repeated accurate measurement;Brain metastases cannot be used as target foci.

  7. Good organ function. 8. The serum pregnancy test results of female subjects in the child-bearing age within 3 days before the first medication were negative; 9. If a fertile female subject has sex with an unsterilized male partner, the subject must begin from screening for effective contraceptive methods and must agree to continue using these precautions until 6 months after the last administration of the study drug;Periodic abstinence, safe period contraception and external ejaculation are not acceptable contraceptive methods.

  10. If an unsterilized male subject has sexual intercourse with a fertile female partner, the subject must use an effective contraceptive method from the beginning of screening to within 6 months after the last dose.

Exclusion Criteria:

* 1. Previous treatment for:Use of small-molecule targeted antitumor drugs, monoclonal or double-clonal antibodies targeting PD-(L)1 or CTLA-4, other anti-tumor antibodies, other anti-tumor therapies (e.g., chemotherapy, radiotherapy, biological or hormonal therapy) within 4 weeks prior to initial administration of the study drug, previous use of immunomodulatory drugs within 2 weeks prior to initial administration of the study drug,Prior treatment with approved or investigational TIGIT antibodies, PVRIG antibodies, or CD96 antibodies.

  2. Enroll in another clinical study at the same time. 3. Received other antitumor therapy 4 weeks before the first administration or 5 half-lives of the drug (whichever is shorter) : e.g. palliative local therapy for non-target lesions was performed within 2 weeks before the first administration;Received non-specific immunomodulatory therapy within 2 weeks prior to initial administration;Received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week prior to initial administration.

  4. Central nervous system metastasis with clinical symptoms. 5. Other malignancies within 3 years prior to the first medication. 6. Active autoimmune disease requiring systemic treatment within 2 years prior to initial medication.

  7. History of serious disease within 1 year before the first medication. 8. History of gastrointestinal perforation and/or fistula, history of gastrointestinal obstruction, and extensive enterectomy within 6 months prior to initial administration.

  9. Patients receiving chest radiotherapy >30 Gy within 6 months before the first drug use, non-chest radiotherapy >30 Gy within 4 weeks before the first drug use, and palliative radiotherapy ≤30 Gy within 2 weeks before the first drug use.Subjects who did not recover from toxicity and/or complications from these interventions to NCI CTCAE grade ≤1 (except hair loss and fatigue).

  10. Live or attenuated vaccine has been administered within 4 weeks prior to initial administration, or if it is planned to be administered during the study period. Inactivated vaccine is permitted .

  11. Severe infection occurs within 4 weeks prior to first dosing. 12. Those who have had major surgical operations or severe trauma within 4 weeks prior to the first dosing, or have major surgical operations planned within 4 weeks after the first dosing; Minor local surgery was performed within 3 days prior to first dosing.

  13. History of severe bleeding tendency or coagulopathy;There were clinically significant bleeding symptoms, including but not limited to gastrointestinal bleeding, hemoptysis, and nasal bleeding, within 4 weeks prior to first dosing .

  14. Systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg after oral antihypertensive medication with present hypertension.

  15. Hyperglycemia that has not been controlled by treatment. 16. Pleural effusion, pericardial effusion or ascites with clinical symptoms or requiring repeated drainage.

  17. There is a history of noninfectious pneumonia requiring systemic glucocorticoid therapy or a current interstitial lung disease.

  18. Active or have a clear history of inflammatory bowel disease. 19.History of immune deficiency; HIV antibody positive; Systemic corticosteroid hormones or other immunosuppressants are currently being used long-term.

  20. Known history of allogeneic organ transplantation and hematopoietic stem cell transplantation.

  21. Untreated subjects with active hepatitis B;Active hepatitis C subjects. 22. No remission of toxicity from previous antitumor therapy, defined as failure to return to the grade 1 level of toxicity defined in NCI, CTCAE 5.0 or below, or the inclusion/exclusion criteria, with the exception of alopecia and fatigue.

  23. Known allergy to any component of any study drug; known history of severe hypersensitivity to other monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events(AE); | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of AK127 and AK104
Incidence of serious adverse events(SAE); | Up to approximately 2 years
  Incidence of SAE is aim to evaluate the safety of AK127 and AK104.
Incidence of immune-related adverse events(irAE); | Up to approximately 2 years
  Incidence of irAE is aim to evaluate the safety of AK127 and AK104.
The incidence of suspected unexpected serious adverse reactions(SUSAR); | Up to approximately 2 years
  The incidence of SUSAR is aim to evaluate the safety of AK127 and AK104.
Incidence of dose-limiting toxicity(DLT); | Up to approximately 2 years
  The purpose of DLT is to find the Phase II recommended dose(RP2D) or MTD.
Number of participants with clinically significant changes in laboratory assessment data as assessed by CTCAE v5.0. | Up to approximately 2 years
  Monitor and summerize all data derive from clinically significant changes in laboratory assessment data per Common Terminology Criteria for Adverse Events(CTCAE)5.0.
AE that leads to the termination or suspension of treatment. | Up to approximately 2 years
  AE that leads to the termination or suspension of treatment is aim to evaluate the safety of AK127 and AK104.

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to approximately 2 years
  ORR is proportion of subjects with complete response(CR) or partial response(PR), based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1(Solid Tumor)or Lugano 2014 Evaluation Criteria(lymphoma).
Disease control rate(DCR) | Up to approximately 2 years
  Disease control rate(DCR) is defined as the proportion of subjects achieving a best of response(BOR) of confirmed CR and PR and stable disease(SD) per RECIST v1.1(Solid Tumor)or Lugano 2014 Evaluation Criteria(lymphoma).
duration of response(DoR) | Up to approximately 2 years
  Duration of response(DoR) is defined as the period from the first documentation of confirmed response(CR or PR) to the first documentation of progressive disease(PD) (as per RECIST v1.1(Solid Tumor)or Lugano 2014 Evaluation Criteria(lymphoma)) or death due to any cause, whichever occurs first.
time to response(TTR) | Up to approximately 2 years
  Time to response(TTR) is defined as the time from the first dose of investigational products until the first confirmation of CR or PR.
progression-free survival(PFS) | Up to approximately 2 years
  Progression-free survival(PFS) is defined as the time from the first dose of investigational products until documentation of progressive disease(PD)(as per RECIST v1.1) or death due to any cause, whichever occurs first.
overall survival(OS) | Up to approximately 2 years
  Overall survival(OS) is defined as the time from the first dose of investigational products until death due to any cause.
The drug concentration of AK127 and AK104 in serum | Up to approximately 2 years
  The drug concentration of AK127 and AK104 in serum was used to assess the blood concentration of AK127 and AK104 at different dosing time points.
maximum concentration(Cmax)of AK127 and AK104 in serum | Up to approximately 2 years
  Maximum concentration(Cmax) is to evaluate the Pharmacokinetics(PK) of AK127 and AK104.
peak time(Tmax) of AK127 and AK104 in serum | Up to approximately 2 years
  Peak time(Tmax)is to evaluate the Pharmacokinetics(PK) of AK127 and AK104.
half time(t1/2) of AK127 and AK104 in serum | Up to approximately 2 years
  Half time(t1/2) is to evaluate the Pharmacokinetics(PK) of AK127 and AK104.
area under curve(AUC)of AK127 and AK104 in serum | Up to approximately 2 years
  Area under curve(AUC) is to evaluate the Pharmacokinetics(PK) of AK127 and AK104.
clearance rate(CL) of AK127 and AK104 in serum | Up to approximately 2 years
  Clearance rate(CL) is to evaluate the Pharmacokinetics(PK) of AK127 and AK104.
apparent volume of distribution(Vd) of AK127 and AK104 in serum | Up to approximately 2 years
  Apparent volume of distribution(Vd) is to evaluate the Pharmacokinetics(PK) of AK127 and AK104.
Number and percentage of subjects with anti-drug antibody(ADA) to AK127 and AK104 | Up to approximately 2 years
  The immunogenicity of AK127 and AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Doctor, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China